CLINICAL TRIAL: NCT06911437
Title: Clinical Study on the Combination of Xiaoyu Zhitong Formula and Lymphatic Drainage Technique to Improve the Symptoms of Knee Pain and Swelling in Cold Dampness Obstruction Type
Status: Enrolling by invitation | Type: Observational
Sponsor: tang jie (Other Government)
Responsible Party: Sponsor-Investigator, tang jie, Director of the Rehabilitation Department of the Hospital of Integrated Traditional Chinese and Western Medicine, Changping District, Beijing, Beijing Municipal Health Commission
Organization: Beijing Municipal Health Commission (Other Government)
Other Study IDs: LunShen(2023)No.09.
Record Dates: First submitted 2025-01-20; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Knee Osteoarthritis (OA)
Keywords: Knee Osteoarthritis; pain; Swelling of soft tissues
MeSH Terms: conditions — Osteoarthritis, Knee; Pain | interventions — Control Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment group: Treatment with Xiaoyu Zhitong Formula combined with lymphatic drainage technique;
  Interventions: Other: treatment group
- Control group: External application of Futalin combined with lymphatic drainage technique for treatment
  Interventions: Other: control group

INTERVENTIONS:
Other: treatment group — Xiaoyu Zhitong Formula: 10g of long pepper, 10g of cloves, 10g of borneol, 10g of papaya, 10g of white peony, 10g of licorice, 15g of chicken blood vine, 10g psoralen, 10g of cistanche, powdered petroleum jelly, wrapped in gauze and heated and applied to the affected area.
  Freehand lymphatic drainage technique: the patient is in the supine position, first use the thumb to press the deep lymph nodes of the trunk for 3-5 min, which are lymph nodes in the groin, neck, lumbosacral spine and supraclavicular fossa, and then perform freehand lymphatic drainage at the lymphatic vessels or superficial lymph nodes, according to the clockwise circle method, all the way to the outside of the thigh, and then to the lateral malleolus of the calf, and then press the medial malleolus of the inner calf to the inner thigh. 20min each time, 1 time every other day. 3 times a week for a total of 9 treatments for 3 weeks.
  Groups: Treatment group
Other: control group — External application of Diclofenac Diethylamine Emulgel（Manufacturer: Switzerland,Haleon CH SARL） combined with lymphatic drainage technique for treatment，Freehand lymphatic drainage technique: the patient is in the supine position, first use the thumb to press the deep lymph nodes of the trunk for 3-5 min, which are lymph nodes in the groin, neck, lumbosacral spine and supraclavicular fossa, and then perform freehand lymphatic drainage at the lymphatic vessels or superficial lymph nodes, according to the clockwise circle method, all the way to the outside of the thigh, and then to the lateral malleolus of the calf, and then press the medial malleolus of the inner calf to the inner thigh. 20min each time, 1 time every other day. 3 times a week for a total of 9 treatments for 3 weeks.
  Groups: Control group

SUMMARY:
This research project applies a combination of blood stasis relieving and pain relieving formula and lymphatic drainage technique to treat patients with cold dampness obstruction type knee joint pain. The improvement of knee joint pain scores and activity function as well as the degree of soft tissue swelling changes are observed before and after receiving this therapy providing certain ideas for the comprehensive treatment optimization and prognosis judgment of cold dampness obstruction type knee joint pain.

ELIGIBILITY:
1. Inclusion Criteria:

   * a. Patients who meet the diagnostic criteria for knee osteoarthritis in the "Guidelines for Diagnosis and Treatment of Osteoarthritis" (2007 edition) of the Chinese Medical Association Orthopedic Branch and also meet the diagnostic criteria for wind cold dampness syndrome of knee joint obstruction;
   * b. Age range: 25-70 years old;
   * c.1 week ≤ disease duration ≤ 2 years;
   * d. If other treatments have already been received and there is a washout period of more than 14 days;
   * e. Voluntarily participate in the study and sign an informed consent form.
2. Exclusion Criteria:

   * a. Patients with bleeding tendencies severe skin damage or skin diseases in certain areas;
   * b. Suspected or diagnosed with tumors;
   * c. Patients with severe heart lung brain diseases tuberculosis osteomyelitis and osteoporosis;
   * d. Patients with mental illnesses;
   * e. Pregnant or planned pregnant women and lactating women;
   * f. Have participated in other clinical studies within the past 3 months;
   * g. The researchers believe that they are not suitable to participate in this clinical study due to other reasons.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with cold dampness obstruction type knee joint pain
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Score | Before treatment and at 1 2 3 and 6 weeks after treatment.
  This method is relatively sensitive and comparable. The specific method is to draw a 10 cm horizontal line on the paper with one end of the line marked as 0 indicating no pain; The other end is 10 indicating severe pain; The middle part represents varying degrees of pain. Ask the patient to draw a mark on the horizontal line based on their own feelings to indicate the degree of pain. The pain score is determined by measuring the length of the mark from the 0 point is the pain score.Quantitative score: A higher score indicates a worse outcome, with 0 being no pain and 10 being the most painful.

SECONDARY OUTCOMES:
Width of soft tissue around joints | Before treatment and at 1, 2, 3, and 6 weeks after treatment.
  Use a tape measure to measure and record at the same position on the knee joint.A lower value indicates a better outcome.
Lysholm knee score scale | Before treatment and at 1, 2, 3, and 6 weeks after treatment.
  Quantitative scoring: Higher scores indicate better outcomes and fewer symptoms or disabilities.
  Qualitative scoring:A score of 95 or above is excellent, 94-85 is good, 84-65 is acceptable, and less than 65 is poor.

CONTACTS AND LOCATIONS:
Locations (1):
- Science and Education Department of Changping District Integrated Traditional Chinese and Western Medicine Hospital Beijing.No. 219 Huangping Road Huoying Changping District Beijing, Beijing, China